CLINICAL TRIAL: NCT02875197
Title: Comparing Running-Specific and Traditional Prostheses During Running: Assessing Performance and Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regis University (Other)
Collaborators: Colorado School of Mines (Unknown)
Responsible Party: Principal Investigator, Brian Baum, Assistant Professor, Regis University
Other Study IDs: OP140064
Record Dates: First submitted 2016-07-14; First posted 2016-08-23 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Amputees; Running With Prosthesis
Keywords: Kinetics; Biomechanics; Amputation; Prosthesis; Transtibial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Controls: Males and females 18-50 years old
  Up to 20 able-bodied sex, age, height, and weight-matched subjects
  Interventions: Other: Running on a treadmill at 6 different speeds
- Lower Extremity Amputees: Males & females 18-50 years old
  * Must have a unilateral, transtibial amputation & must have been prescribed a running-specific prosthesis
  * Subject with amputations resulting from trauma, congenital reasons, or cancer treatment unless cancer is in remission or treatments do not impact gait function
  * Physician approval to run
  * 4 months experience using a running-specific prosthesis
  Interventions: Other: Running on a treadmill at 6 different speeds

INTERVENTIONS:
Other: Running on a treadmill at 6 different speeds — All subjects will be required to run at 6 prescribed speeds (2.5, 3.0, 3.5, 4.0, 5.0, and 6.0 m/sec) on a treadmill completing at least 10 consecutive strides, or running for 30 seconds.

SUMMARY:
The purpose of this research is to provide clinically, administratively, and field-relevant objective running outcomes by directly comparing running biomechanics of individuals with lower extremity amputation (ILEA) using RSPs (Running Specific Prostheses) and traditional prostheses. Within this purpose, the project has two specific aims:

Specific Aim 1: To compare RSPs and traditional prostheses with respect to running ability and performance

Specific Aim 2: To compare RSPs and traditional prostheses with respect to injury risks associated with running

Hypothesis 1a: RSPs will outperform traditional prostheses at all velocities as measured by kinetic data (ground reaction forces, joint powers, joint and limb work) and 50m dash time.

Hypothesis 1b: ILEA intact limbs and able-bodied control limbs will outperform residual limbs with RSPs and traditional prostheses at all velocities as measured by kinetic data.

Hypothesis 2: Running with RSPs will show reduced acute and chronic injury risks compared to traditional prostheses at all velocities as measured by loading rates, EMG amplitudes, lumbopelvic kinematics, and modeled joint loads.

DETAILED DESCRIPTION:
A. BACKGROUIND

Current knowledge and understanding of individuals with lower extremity amputations (ILEA) when running are limited with respect to biomechanical performance and injury risks. ILEA are able to run with both running-specific prostheses (RSPs) and traditional prostheses; however, direct comparisons of subjects running with each of these prosthetic designs do not exist. The reported literature examining one design or the other often do not have participants running at the same velocities. Additionally, when running velocities are similar between studies, the same variables are rarely investigated. This makes comparisons between RSPs and traditional prostheses exceedingly difficult, and drawing conclusions on both performance and injury risk is virtually impossible. Furthermore, no ILEA running studies to date have investigated muscle activities, nor have running simulations of musculoskeletal models been generated. These major gaps in research substantially limit the understanding of both performance and injury risk of ILEA running with different prosthetic designs. Gaining this knowledge will directly inform clinicians and administrators within the Department of Defense and Veterans Administration systems on prosthesis prescription for running at a range of speeds as well as for return to duty scenarios. Therefore, the proposed study will utilize motion capture, muscle activity, and musculoskeletal modeling techniques to directly compare performance and injury risks of ILEA running with both RSPs and traditional prostheses across a range of speeds. The investigators will also capture an able-bodied control group for normative comparisons. In doing so, this project directly attends to the OPORA's goals and needs at multiple levels.

B. RESEARCH STRATEGY:

Subjects Twelve subjects with unilateral transtibial amputations will be recruited from the military, veteran, and civilian populations. Twelve able-bodied sex, age, height, and weight-matched subjects will serve as a control group to provide normative data for comparison. All subjects must provide their informed consent prior to beginning any portion of the study and will have the option to discontinue the study at any time without penalty. All subjects must complete the Physical Activity Readiness Questionnaire (PAR-Q) prior to beginning the experiment. If subjects fail this questionnaire (by responding "yes" to any of the 7 questions), they will not be allowed to participate in the study until they provide documentation from a physician clearing them to participate.

Experimental Procedures A randomization computer program will determine the order of prosthetic foot conditions (RSP or traditional) for the ILEA subjects. All subjects (Controls and ILEA) will undergo 3D running analysis on an instrumented treadmill. A motion capture system will collect kinematic data (i.e. limb positions; joint angles, velocities, accelerations) at 200 Hz from reflective markers placed on specific body landmarks. On the amputated limb, the shank cluster will be placed laterally on the socket and a marker will be placed at the distal tip of the socket to define the long axis of the residual shank segment. For the RSP conditions, eight additional markers will be placed on the prosthesis keel. The marker on the most acute point of the prosthesis will define the prosthetic limb "ankle" joint. For the traditional prosthesis conditions, markers will be placed similarly to the intact foot.

An instrumented treadmill will collect ground reaction force (GRF) data at 1000 Hz from force platforms imbedded in the treadmill. Kinematic and ground reaction force data will be combined and standard inverse dynamics techniques will be used to calculate joint kinetic data (i.e. forces, moments, powers, and work) using Visual3D (C-Motion, Germantown, MD) software.

Muscle activation data will be collected at a sampling frequency of 2000 Hz using surface electromyography (EMG) from six bilateral hip and trunk muscles. Disposable pre-gelled silver-silver chloride (Ag-AgCl) electrodes will be placed over bilateral gluteus medius, gluteus maximus, rectus femoris, biceps femoris, lumbar erector spinae, internal oblique, and external oblique muscles. Maximal voluntary isometric contractions (MVIC) will be obtained for normalization purposes using manual resistance applied in standardized positions.

All subjects (ILEA using RSPs, ILEA using traditional prosthesis, and Controls) will run at six prescribed speeds (2.5, 3.0, 3.5, 4.0, 5.0, 6.0 m/s) on a treadmill, presented in randomized order. ILEA subjects will complete all speed conditions wearing both their RSP and traditional prosthetic foot. As mentioned earlier, the prosthesis order will be randomized, but all speed conditions will be completed in one prosthesis prior to changing into the second prosthesis condition. This will save time and maintain a similar prosthetic fit between speed conditions. The study protocol requires that every subject runs at the same 6 specific speeds identified above. Each treadmill speed condition will take approximately 30 seconds, or the time needed for subjects to stabilize their gait at the speed and a collection of 10 consecutive strides to be collected. At least 2 minutes rest will be provided between each speed condition, and subjects can take more rest if needed.

After completing the treadmill trials, subjects will complete 3x50m dashes in each foot condition to determine maximum speed. Again, at least 2 minutes rest will be provided between each effort, and subjects can take more rest if needed. The order of prosthesis use will also be randomized for this test, but all three dashes will be completed consecutively for each prosthesis condition.

To evaluate performance while running, the primary outcome measures being evaluated will include peak joint powers; concentric, eccentric and total joint and limb work; average vertical and Anterior and Posterior (AP) GRFs; vertical and AP GRF impulses; and 50m dash time/speed. To evaluate injury risk while running, the primary outcome measures being evaluated will include average GRF magnitudes and loading rates, asymmetry in GRFs and joint moments, normalized EMG amplitudes, lumbopelvic kinematics, and peak and average joint contact forces over stance. Data for these measures will be collected for all subjects and then compared among the three groups (ILEA with RSPs, ILEA with Traditional Prosthesis, and Controls). No intervention will be offered to any subject and no follow-up to assess biomedical and/or health outcomes will be conducted.

Electromyography Signal Analysis Raw EMG data will be demeaned, band-pass (cutoff frequency10-400 Hz) and band-stop (cutoff frequency 59-61 Hz) filtered to remove movement artifact and 60 Hz electrical noise using dual-pass (zero phase lag) Butterworth filters. EMG data will then be full wave rectified and low pass filtered to create linear envelopes. Peak values will be extracted from the MVIC trials to be used for normalization of the running trials to express EMG data as % Maximum Voluntary Contraction (MVC). Root mean square (RMS) of each muscle's activity will be calculated during stance and swing phases of running to investigate amplitude differences. Cross-correlation methodology will be utilized to investigate relative timing between trunk and hip musculature. Comparisons will be made to assess symmetry of muscle activation amplitude and timing between intact and prosthetic limb sides for each of the running speed and prosthesis conditions.

Musculoskeletal Model Three musculoskeletal models will be developed in OpenSim. For the first model, the investigators will use a generic musculoskeletal model representing a non-amputee adult male, which has previously been used to assess muscle function during non-amputee running. The second and third models will be modified versions of the non-amputee model that represents a person using a prosthesis. The second model will include a traditional transtibial energy storage and return prosthesis, and the third model will include a running specific prosthesis. For both models, the investigators will remove the ankle muscles from the residual leg, including the medial and lateral gastrocnemius, soleus, tibialis posterior, flexor digitorum longus, tibialis anterior and extensor digitorum longus.

Running Simulation Generation The models will be scaled to each individual subject using manual, uniform scale factors, computed from an inverse dynamics model based on kinematic marker positions and developed in Visual3D (C-Motion, Inc., Germantown, MD). Then, an inverse kinematics solution will be computed in Visual3D using a weighted least squares optimization algorithm. After the inverse kinematics solution has been computed, the investigators will perform a Residual Reduction Algorithm. Once minor changes have been made to the model and to the kinematic trajectories of the generalized coordinates, the investigators will implement a Computed Muscle Control algorithm. Once a solution for individual muscle excitations is found using the Computed Muscle Control algorithm, the investigators will compare it to the experimentally-collected electromyographic data. The investigators will generate running simulations at all running speeds for all participants. The results of these simulations will be compared between groups and across speeds, similar to the experimental measures that will be analyzed in this study.

Joint Contact Force Analysis Once the running simulations have been developed, the three-dimensional contact load at the hip will be determined from the joint intersegmental force and compressive forces from the muscles crossing the joint, similar to the previous analyses during amputee walking. In addition, the muscle forces determined from the movement simulation will be used to help interpret the net contact loads.

Material Properties and Anthropometrics Inertial properties of the prosthetic components and intact body segments will be estimated for use with the inverse dynamics approach. Subject masses will be measured using a force platform. Height and body weight of each subject will be measured, and anthropometric measurements from marker positions will be used to estimate the mass, center of mass, and moments of inertia of intact limb segments. Because ILEA subjects are missing one foot and part of their shank, an adjusted body mass (ABM) will be used as an input to anthropometric regression equations that account for the missing body segments.

For subjects with amputation, the residual limb length and circumferences at the knee joint and distal end of the limb will be measured using a measuring tape. Residual limb inertial properties will then be estimated as a frustum of a right circular cone. Residual limb mass will be estimated from the calculated geometric volume assuming a uniform 1.10 g/cm3 tissue density. For the RSP conditions, the inertial properties of the RSP will be estimated from data published by the PI. Subsegments within the RSP keels will be defined via reflective marker placements and the inertial properties of each subsegment will be estimated by assuming each segment as a rigid trapezoidal cuboid. For the traditional prosthesis conditions, the inertial properties of the prosthesis will be estimated according to published literature.

C. STATISTICAL PLAN and DATA ANALYSIS

Statistical Analysis This research is designed to determine the effects of prosthesis type on a variety of performance and injury-risk related outcome variables across a range of running speeds. A three factor (Group x Limb x Speed) mixed model ANOVA will be used to identify statistical changes of the following dependent variables: peak hip, knee, and ankle joint powers and mechanical work; average ground reaction forces; loading rates; and EMG amplitudes. Group (Individual Lower Extremity Amputation Running-Specific Prosthesis (ILEARSP) vs Individual Lower Extremity Amputation Traditional Prosthesis (ILEATrad) vs. Control) will be considered as a between-subjects independent variable, Limb (prosthetic/intact or left/right) as a within-subjects independent variable and Speed (2.5, 3.0, 3.5, 4.0, 5.0, and 6.0 m/s) as a within-subjects independent variable.

A two factor (Group x Speed) ANOVA will be used to identify statistical changes of dependent variables including ground reaction force symmetry, joint kinetic symmetry, and lumbopelvic kinematics. A one-way ANOVA will determine statistical differences between groups for the 50m dash time and speed.

Significance for all statistical tests will be set at α=0.05.

Sample Size Calculations This study will have appropriate statistical power to assess our hypotheses. Effect sizes for significant differences between RSP, intact, and able-bodied limbs in GRF loading rates, average GRF, and total joint work were estimated based on prior data collected by the PI from 8 ILEA and Control subjects running at 2.5, 3.0, and 3.5 m/s. These effect sizes ranged between 0.4 and greater than 0.9. An effect size of 0.7 was also estimated from the volume of oxygen (VO2) values of one study comparing subjects running with RSPs and traditional prostheses. To be conservative, the investigators utilized the lowest of these effect sizes (0.4) to perform a power analysis for ANOVA with repeated measures using G*Power (v. 3.1.9.2, Dusseldorf, Germany). This yielded a total sample size of 24 with α = 0.05 resulting in 80% power to detect differences between limbs, prosthetic feet, or ILEA and Control subjects in kinetic values during running. The investigators anticipate similar effect sizes for changes in the remaining biomechanical variables the investigators will examine in the proposed study. Based on this analysis, 12 ILEA subjects and 12 control subjects will provide substantial statistical power to detect significant differences in biomechanical outcomes between groups and prosthetic feet.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with amputation must have a unilateral, transtibial amputation and must have been prescribed a running-specific prosthesis
* Subject with amputations resulting from trauma, congenital reasons, or cancer treatment. If due to cancer, cancer must be in remission or subjects must not be undergoing treatments that could affect their gait function
* Subjects with amputation must be cleared to run by a physician
* Subjects with amputation must have at least 4 months experience using a running-specific prosthesis
* All subjects must be between the ages of 18 and 50 years
* Males and females who meet the inclusion/exclusion criteria are eligible to participate

Exclusion Criteria:

* Subjects with any injury, affliction, or comorbidities to the limb(s) (other than the amputation) that impairs the gait pattern
* Women who are pregnant, as pregnancy can affect the gait pattern
* Amputations resulting from dysvascular disease as this may affect their gait function
* Amputations resulting from cancer treatment where the subject is still undergoing treatment that may affect their gait function

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Up to twenty subjects with unilateral transtibial amputations will be recruited from the military, veteran, and civilian populations. Civilian individuals with lower extremity amputation (ILEA) will be recruited who match the age range of military service members commonly sustaining injuries resulting in amputation. Up to twenty able-bodied sex, age, height, and weight-matched subjects will serve as a control group to provide normative data for comparison.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Peak Joint Powers | Assessed on day 1 (data collection day)
  Peak joint power, calculated as the product of joint torque and joint angular velocity, is the highest power value achieved during the movement being evaluated and is measured in watts or watts per kg if normalized based on body weight.
Concentric, Eccentric, and Total Joint and Limb Work. | Assessed on day 1 (data collection day)
  Concentric, eccentric, and total joint and limb work is defined as force multiplied by displacement, and is expressed in watts.
Average Ground Reaction Forces. | Assessed on day 1 (data collection day)
  Ground reaction force is the equaling and opposing force due to body mass passing through the foot to the ground surface; ground reaction forces is resolved into vertical (counteracting body weight) and horizontal (anterior and posterior) components. Ground reaction forces are expressed in newtons.
Ground Reaction Force Impulses | Assessed on day 1 (data collection day)
  Vertical and anteroposterior ground reaction force impulses are determined by multiplying the impact force by the time over which the impact force acts. Impulses are stated in newton-seconds.
Average Ground Reaction Force Magnitudes | Assessed on day 1 (data collection day)
  Ground reaction forces is defined as the force exerted by the ground on the body in contact with the ground. Ground reaction force magnitudes will be averaged and expressed in newtons.
Average Ground Reaction Force Loading Rates | Assessed on day 1 (data collection day)
  Ground reaction force loading rate is the speed at which forces impact the body, and is calculated by dividing the maximal vertical force by the time needed to reach the maximal vertical force. It is expressed in body weights per millisecond.
Ground Reaction Forces | Assessed on day 1 (data collection day)
  Asymmetry in ground reaction forces and joint moments is determined by statistical differences between the left and right side.
Normalized EMG Amplitudes | Assessed on day 1 (data collection day)
  EMG amplitudes will be measured in millivolts and then normalized based on EMG amplitudes measured during maximum voluntary contractions using a scale of 0 to 1.
Lumbopelvic Kinematics | Assessed on day 1 (data collection day)
  Lumbopelvic kinematics is a postural evaluation of the lumbopelvic region expressing positions in degrees or radians.
Joint Contact Forces over Stance | Assessed on day 1 (data collection day)
  Peak and average joint contact forces are forces that occur over stance (while there is contact between a limb and the ground). Peak forces are the highest force that occurs during stance, while average forces is the average of all force levels occuring during stance. Force measurements are expressed in newtons.
50 Meter Dash | Assessed on day 1 (data collection day)
  A 50 meter dash effort will be used as an indicator of maximum running speed. It will be reported as an average of three trials and expressed as total time in seconds and as speed expressed in meters per second.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Baum, Ph.D., Principal Investigator — Assistant Professor
Locations (1):
- Regis University, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bussmann JB, Grootscholten EA, Stam HJ. Daily physical activity and heart rate response in people with a unilateral transtibial amputation for vascular disease. Arch Phys Med Rehabil. 2004 Feb;85(2):240-4. doi: 10.1016/s0003-9993(03)00485-4. PMID 14966708
- [Result] Naschitz JE, Lenger R. Why traumatic leg amputees are at increased risk for cardiovascular diseases. QJM. 2008 Apr;101(4):251-9. doi: 10.1093/qjmed/hcm131. Epub 2008 Feb 16. PMID 18281705
- [Result] Saris WH, Blair SN, van Baak MA, Eaton SB, Davies PS, Di Pietro L, Fogelholm M, Rissanen A, Schoeller D, Swinburn B, Tremblay A, Westerterp KR, Wyatt H. How much physical activity is enough to prevent unhealthy weight gain? Outcome of the IASO 1st Stock Conference and consensus statement. Obes Rev. 2003 May;4(2):101-14. doi: 10.1046/j.1467-789x.2003.00101.x. PMID 12760445
- [Result] Singh R, Hunter J, Philip A. The rapid resolution of depression and anxiety symptoms after lower limb amputation. Clin Rehabil. 2007 Aug;21(8):754-9. doi: 10.1177/0269215507077361. PMID 17846075
- [Result] Yap TL, Davis LS. Physical activity: the science of health promotion through tailored messages. Rehabil Nurs. 2008 Mar-Apr;33(2):55-62. doi: 10.1002/j.2048-7940.2008.tb00204.x. PMID 18330383
- [Result] Poirier P, Despres JP. Exercise in weight management of obesity. Cardiol Clin. 2001 Aug;19(3):459-70. doi: 10.1016/s0733-8651(05)70229-0. PMID 11570117
- [Result] Kavanagh T. Exercise and the heart. Ann Acad Med Singap. 1983 Jul;12(3):331-7. PMID 6378048
- [Result] Kram R, Grabowski AM, McGowan CP, Brown MB, Herr HM. Counterpoint: Artificial legs do not make artificially fast running speeds possible. J Appl Physiol (1985). 2010 Apr;108(4):1012-4; discussion 1014; author reply 1020. doi: 10.1152/japplphysiol.01238.2009a. No abstract available. PMID 20368386
- [Result] Weyand PG, Bundle MW. Point: Artificial limbs do make artificially fast running speeds possible. J Appl Physiol (1985). 2010 Apr;108(4):1011-2; discussion 1014-5. doi: 10.1152/japplphysiol.01238.2009. No abstract available. PMID 20368385
- [Result] Brown MB, Millard-Stafford ML, Allison AR. Running-specific prostheses permit energy cost similar to nonamputees. Med Sci Sports Exerc. 2009 May;41(5):1080-7. doi: 10.1249/MSS.0b013e3181923cee. PMID 19346979
- [Result] Baum BS. Kinetics in individuals with unilateral transtibial amputations using running-specific prostheses, Dissertation, University of Maryland, College Park, Md., 2012.
- [Result] Grabowski AM, McGowan CP, McDermott WJ, Beale MT, Kram R, Herr HM. Running-specific prostheses limit ground-force during sprinting. Biol Lett. 2010 Apr 23;6(2):201-4. doi: 10.1098/rsbl.2009.0729. Epub 2009 Nov 4. PMID 19889694
- [Result] Sanderson DJ, Martin PE. Joint kinetics in unilateral below-knee amputee patients during running. Arch Phys Med Rehabil. 1996 Dec;77(12):1279-85. doi: 10.1016/s0003-9993(96)90193-8. PMID 8976312
- [Result] Czerniecki JM, Gitter A. Insights into amputee running. A muscle work analysis. Am J Phys Med Rehabil. 1992 Aug;71(4):209-18. doi: 10.1097/00002060-199208000-00003. PMID 1642820
- [Result] Czerniecki JM, Gitter A, Munro C. Joint moment and muscle power output characteristics of below knee amputees during running: the influence of energy storing prosthetic feet. J Biomech. 1991;24(1):63-75. doi: 10.1016/0021-9290(91)90327-j. PMID 2026634
- [Result] Czerniecki JM, Gitter AJ, Beck JC. Energy transfer mechanisms as a compensatory strategy in below knee amputee runners. J Biomech. 1996 Jun;29(6):717-22. doi: 10.1016/0021-9290(95)00173-5. PMID 9147968
- [Result] Buckley JG. Biomechanical adaptations of transtibial amputee sprinting in athletes using dedicated prostheses. Clin Biomech (Bristol). 2000 Jun;15(5):352-8. doi: 10.1016/s0268-0033(99)00094-7. PMID 10758296
- [Result] Heiderscheit BC, Chumanov ES, Michalski MP, Wille CM, Ryan MB. Effects of step rate manipulation on joint mechanics during running. Med Sci Sports Exerc. 2011 Feb;43(2):296-302. doi: 10.1249/MSS.0b013e3181ebedf4. PMID 20581720
- [Result] Novacheck TF. The biomechanics of running. Gait Posture. 1998 Jan 1;7(1):77-95. doi: 10.1016/s0966-6362(97)00038-6. PMID 10200378
- [Result] Winter DA. Moments of force and mechanical power in jogging. J Biomech. 1983;16(1):91-7. doi: 10.1016/0021-9290(83)90050-7. No abstract available. PMID 6833314
- [Result] Nyland J, Snouse SL, Anderson M, Kelly T, Sterling JC. Soft tissue injuries to USA paralympians at the 1996 summer games. Arch Phys Med Rehabil. 2000 Mar;81(3):368-73. doi: 10.1016/s0003-9993(00)90086-8. PMID 10724085
- [Result] Ferrara MS, Peterson CL. Injuries to athletes with disabilities: identifying injury patterns. Sports Med. 2000 Aug;30(2):137-43. doi: 10.2165/00007256-200030020-00006. PMID 10966152
- [Result] Crowell HP, Davis IS. Gait retraining to reduce lower extremity loading in runners. Clin Biomech (Bristol). 2011 Jan;26(1):78-83. doi: 10.1016/j.clinbiomech.2010.09.003. PMID 20888675
- [Result] Williams KR, Cavanagh PR, Ziff JL. Biomechanical studies of elite female distance runners. Int J Sports Med. 1987 Nov;8 Suppl 2:107-18. doi: 10.1055/s-2008-1025715. PMID 3692651
- [Result] Miller DI. Resultant lower extremity joint moments in below-knee amputees during running stance. J Biomech. 1987;20(5):529-41. doi: 10.1016/0021-9290(87)90253-3. PMID 3611127
- [Result] McGowan CP, Grabowski AM, McDermott WJ, Herr HM, Kram R. Leg stiffness of sprinters using running-specific prostheses. J R Soc Interface. 2012 Aug 7;9(73):1975-82. doi: 10.1098/rsif.2011.0877. Epub 2012 Feb 15. PMID 22337629
- [Result] Hobara H, Baum BS, Kwon HJ, Linberg A, Wolf EJ, Miller RH, Shim JK. Amputee locomotion: lower extremity loading using running-specific prostheses. Gait Posture. 2014;39(1):386-90. doi: 10.1016/j.gaitpost.2013.08.010. Epub 2013 Aug 18. PMID 24035367
- [Result] Milner CE, Ferber R, Pollard CD, Hamill J, Davis IS. Biomechanical factors associated with tibial stress fracture in female runners. Med Sci Sports Exerc. 2006 Feb;38(2):323-8. doi: 10.1249/01.mss.0000183477.75808.92. PMID 16531902
- [Result] Zadpoor AA, Nikooyan AA. The relationship between lower-extremity stress fractures and the ground reaction force: a systematic review. Clin Biomech (Bristol). 2011 Jan;26(1):23-8. doi: 10.1016/j.clinbiomech.2010.08.005. Epub 2010 Sep 16. PMID 20846765
- [Result] Waetjen L, Parker M, Wilken JM. The effects of altering initial ground contact in the running gait of an individual with transtibial amputation. Prosthet Orthot Int. 2012 Sep;36(3):356-60. doi: 10.1177/0309364611433353. PMID 22918914
- [Result] Burkett B, Smeathers J, Barker T. Walking and running inter-limb asymmetry for Paralympic trans-femoral amputees, a biomechanical analysis. Prosthet Orthot Int. 2003 Apr;27(1):36-47. doi: 10.3109/03093640309167975. PMID 12812326
- [Result] Buckley JG. Sprint kinematics of athletes with lower-limb amputations. Arch Phys Med Rehabil. 1999 May;80(5):501-8. doi: 10.1016/s0003-9993(99)90189-2. PMID 10326911
- [Result] Collins JJ, Whittle MW. Influence of gait parameters on the loading of the lower limb. J Biomed Eng. 1989 Sep;11(5):409-12. doi: 10.1016/0141-5425(89)90105-2. PMID 2796321
- [Result] Keller TS, Weisberger AM, Ray JL, Hasan SS, Shiavi RG, Spengler DM. Relationship between vertical ground reaction force and speed during walking, slow jogging, and running. Clin Biomech (Bristol). 1996 Jul;11(5):253-259. doi: 10.1016/0268-0033(95)00068-2. PMID 11415629
- [Result] Munro CF, Miller DI, Fuglevand AJ. Ground reaction forces in running: a reexamination. J Biomech. 1987;20(2):147-55. doi: 10.1016/0021-9290(87)90306-x. PMID 3571295
- [Result] Nilsson J, Thorstensson A. Ground reaction forces at different speeds of human walking and running. Acta Physiol Scand. 1989 Jun;136(2):217-27. doi: 10.1111/j.1748-1716.1989.tb08655.x. PMID 2782094
- [Result] Silverman AK, Fey NP, Portillo A, Walden JG, Bosker G, Neptune RR. Compensatory mechanisms in below-knee amputee gait in response to increasing steady-state walking speeds. Gait Posture. 2008 Nov;28(4):602-9. doi: 10.1016/j.gaitpost.2008.04.005. Epub 2008 Jun 2. PMID 18514526
- [Result] Isakov E, Burger H, Krajnik J, Gregoric M, Marincek C. Knee muscle activity during ambulation of trans-tibial amputees. J Rehabil Med. 2001 Sep;33(5):196-9. doi: 10.1080/165019701750419572. PMID 11585149
- [Result] Fey NP, Klute GK, Neptune RR. The influence of energy storage and return foot stiffness on walking mechanics and muscle activity in below-knee amputees. Clin Biomech (Bristol). 2011 Dec;26(10):1025-32. doi: 10.1016/j.clinbiomech.2011.06.007. Epub 2011 Jul 20. PMID 21777999
- [Result] Ventura JD, Klute GK, Neptune RR. The effect of prosthetic ankle energy storage and return properties on muscle activity in below-knee amputee walking. Gait Posture. 2011 Feb;33(2):220-6. doi: 10.1016/j.gaitpost.2010.11.009. Epub 2010 Dec 9. PMID 21145747
- [Result] Brüggemann GP, Arampatzis A, Emrich F, Potthast W. Biomechanics of double transtibial amputee sprinting using dedicated sprinting prostheses. Sports Technol 1: 220-227, 2009.
- [Result] Feldman DR, Gonzalez-Fernandez M, Singla AA, Krabak BJ, Singh S, Krabak J, Singh S. Hip and pelvis injuries in special populations, in: Seidenberg P, Bowen JD. (Eds.), The Intact Hip and Pelvis in Sports Medicine and Primary Care. Springer, New York, 187-205, 2010.
- [Result] Laboute E, Druvert JC, Pailler D, Piera JB. [Stress fractures in disabled athletes' preparation for the paralympic games in Athens, 2004: an assessment]. Ann Readapt Med Phys. 2008 Mar;51(2):114-8. doi: 10.1016/j.annrmp.2007.12.001. Epub 2008 Jan 7. French. PMID 18241949
- [Result] Hobara H, Baum BS, Kwon HJ, Shim JK. Running mechanics in amputee runners using running-specific prostheses. Jap J Biomech Sports Exerc 17: 53-61, 2013.
- [Result] Zatsiorsky VM. Kinetics of Human Motion. Human Kinetics. Champaign, IL, 2002.
- [Result] Zipp P. Recommendations for the standardization of lead positions in surface electromyography. Eur J Appl Physiol Occup Physiol 50: 41-54, 1982.
- [Result] Kendall FP, McCreary EK, Provance PG, Rodgers MM, Romani WA. Muscles: Testing and Function, with Posture and Pain, 5th ed. Lippincott Williams & Wilkins, Baltimore, MD, 2005.
- [Result] Winter DA. Biomechanics and Motor Control of Human Movement. John Wiley & Sons, Hoboken, NJ, 2009.
- [Result] Smith JD. Effects of prosthesis inertia on the mechanics and energetics of amputee locomotion. Dissertation. The Pennsylvania State University, 2008.
- [Result] Mattes SJ, Martin PE, Royer TD. Walking symmetry and energy cost in persons with unilateral transtibial amputations: matching prosthetic and intact limb inertial properties. Arch Phys Med Rehabil. 2000 May;81(5):561-8. doi: 10.1016/s0003-9993(00)90035-2. PMID 10807092